CLINICAL TRIAL: NCT01475175
Title: Adaptive Cardiac Resynchronization Therapy Optimization at Rest and During Exercise (AdOPT CRT)
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to reach sample size to satisfy the primary objective
Sponsor: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AdOPT CRT Sub Study
Record Dates: First submitted 2011-11-16; First posted 2011-11-21 (Estimated); Results first posted 2012-10-12 (Estimated); Last update posted 2019-08-05 (Actual); Status verified 2019-06

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

ARMS (1):
- CRT pacing at rest and during exercise (Experimental): Rest and sub-maximal exercise
  Interventions: Device: CRT pacing at rest and during exercise

INTERVENTIONS:
Device: CRT pacing at rest and during exercise — CRT pacing with aCRT settings and BiV pacing with nominal programming at rest and during submaximal exercise

SUMMARY:
The AdOPT Cardiac Resynchronization Therapy (CRT) study is an acute, prospective, multi-center, non-randomized investigational study designed to compare indices of cardiac function at device settings optimized using the investigational Adaptive CRT (aCRT) algorithm versus nominal programming. The comparison will be performed during rest, atrial pacing and sub-maximal exercise. AdOPT CRT is a sub study of the Adaptive CRT Study (NTC00980057) being conducted in Europe.

DETAILED DESCRIPTION:
Adaptive CRT is an implantable heart failure device feature that attempts to optimize CRT without echocardiographic testing.

ELIGIBILITY:
Inclusion Criteria:

* Subject is age 18 or greater
* Subject is willing to sign and date the study Informed Consent form
* Subject has been implanted with a clinically indicated CRT-D device (Medtronic Vision 3D or Protecta models) for at least 1 month but less than 7 months from the date of study enrollment

Exclusion Criteria:

* Subject has a history of persistent or permanent AF for which pharmacological therapy and/or cardioversion have been unsuccessful or have not been attempted.
* Subject has atrial or ventricular tachyarrhythmias or frequent atrial or ventricular ectopy at the time of enrollment.
* Subject's resting heart rate at the time of enrollment exceeds 90 bpm.
* Subject had CRT system implanted for more than 7 months from the date of the study enrollment
* Subject has complete AV block.
* Subject had previous mechanical valve surgeries.
* Subject has congenital heart disease.
* Subject has contraindication for an exercise test.
* Subject is unable to perform a sub-maximal exercise test.
* It is not possible to acquire technically acceptable echocardiographic images.
* Subject has medical conditions that would limit study participation.
* Subject is pregnant (all women of child-bearing potential must undergo a pregnancy test within seven days prior to the study visit).
* Subject is enrolled in the Adaptive CRT study
* Subject is enrolled in concurrent studies which could confound the results of this study.
* Subject meets exclusion criteria required by local law

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2011-11 (Actual); Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: AdOPT CRT/aCRT Study Team, Study Chair — Medtronic
Locations (7):
- Linz, Austria
- Belgium (2):
  - Genk
  - Leuven
- Aarhus, Denmark
- Lüdenscheid, Germany
- Nijmegen, Netherlands
- Oslo, Norway

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Twelve subjects were enrolled at six centers in Europe between November 2011 and March 2012.
Groups:
- Adaptive CRT Pacing: Cardiac resynchronization therapy (CRT) with adaptive pacing.
Period: Overall Study
Arm/Group | Adaptive CRT Pacing
Started | 12
Completed | 12
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Adaptive CRT Pacing
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 7
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.3 (16.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 10
Region of Enrollment [Number; unit: participants]
  Belgium | 2
  Denmark | 1
  Austria | 2
  Norway | 2
  Netherlands | 3
  Germany | 2

OUTCOME MEASURES:

1. Primary Outcome: Stroke Volume at Rest
Description: Difference in stroke volume (SV) between BiV pacing with aCRT settings and BiV pacing with nominal settings at rest. Biventricular pacing is a type of pacing that paces both the right and left ventricles of the heart. Stroke volume is the volume of blood pumped from a ventricle in one heart beat.
Time Frame: Test day visit (within 14 days of enrollment)
Population: Echo SV data was complete for all 12 subjects.Two patients were programmed incorrectly during the study procedure.
Measure: Mean (95% Confidence Interval); unit: mL
Arm/Group | Adaptive CRT Pacing
Number analyzed (Participants) | 10
mL | 12.1 [8.4 to 22.2]

2. Primary Outcome: Stroke Volume During Atrial Pacing.
Description: Difference in SV between BiV pacing with aCRT settings and BiV pacing with nominal settings during atrial pacing. Atrial pacing occurs at 20 beats-per-minute (bpm) above the subject's resting heart rate.
Time Frame: Test day visit (within 14 days of enrollment)
Population: Echo SV data was complete for all 12 subjects.
Measure: Mean (95% Confidence Interval); unit: mL
Arm/Group | Adaptive CRT Pacing
Number analyzed (Participants) | 12
mL | 9.4 [6.7 to 16]

3. Primary Outcome: Stroke Volume During Sub-maximal Exercise.
Description: Difference in SV between BiV pacing with aCRT settings and BiV pacing with nominal settings during sub-maximal exercise. Sub-maximal exercise is exercise performed at a level below maximum effort. The subject will perform sub-maximal exercise to achieve target heart rate close to 75% of the age-predicted maximal heart rate.
Time Frame: Test day visit (within 14 days of enrollment)
Population: Echo SV data was complete for all 12 subjects.
Measure: Mean (95% Confidence Interval); unit: mL
Arm/Group | Adaptive CRT Pacing
Number analyzed (Participants) | 12
mL | 11.3 [8.0 to 19.2]

4. Secondary Outcome: Cardiac Function With aCRT Settings at Rest
Description: Difference in blood pressure (BP)-derived and echocardiogram (echo)-derived parameters of cardiac function between BiV pacing with aCRT settings and BiV pacing with nominal settings at rest.
Time Frame: Test day visit (within 14 days of enrollment)
Population: Data were not collected.
Arm/Group | Adaptive CRT Pacing
Number analyzed (Participants) | 0

5. Secondary Outcome: Cardiac Function With Nominal Settings at Rest.
Description: Difference in BP-derived and echo-derived parameters of cardiac function between BiV pacing with nominal settings and intrinsic conduction at rest.
Time Frame: Test day visit (within 14 days of enrollment)
Population: Data were not collected
Arm/Group | Adaptive CRT Pacing
Number analyzed (Participants) | 0

6. Secondary Outcome: Cardiac Function With aCRT Settings During Sub-maximal Exercise.
Description: Difference in BP-derived and echocardiogram (echo)-derived parameters of cardiac function between BiV pacing with aCRT settings and BiV pacing with nominal settings during sub-maximal exercise.
Time Frame: Test day visit (within 14 days of enrollment)
Population: Data were not collected.
Arm/Group | Adaptive CRT Pacing
Number analyzed (Participants) | 0

7. Secondary Outcome: Cardiac Function With Nominal Settings During Sub-maximal Exercise.
Description: Difference in BP-derived and echo-derived parameters of cardiac function between BiV pacing with nominal settings and intrinsic conduction during sub-maximal exercise.
Time Frame: Test day visit (within 14 days of enrollment)
Population: Data were not collected.
Arm/Group | Adaptive CRT Pacing
Number analyzed (Participants) | 0

8. Secondary Outcome: Electrical Conduction at Rest.
Description: Electrical conduction will be evaluated at rest by measuring the subject's intrinsic atrio-ventricular (AV) interval. The AV interval is the amount time between the start of atrial contraction and the start of ventricular contraction.
Time Frame: Test day visit (within 14 days of enrollment)
Population: Data were not collected.
Arm/Group | Adaptive CRT Pacing
Number analyzed (Participants) | 0

9. Secondary Outcome: Electrical Conduction During Sub-maximal Exercise.
Description: Electrical conduction will be evaluated during sub-maximal exercise by measuring the subject's intrinsic AV interval.
Time Frame: Time Frame: Test day visit (within 14 days of enrollment)
Population: Data were not collected.
Arm/Group | Adaptive CRT Pacing
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Adaptive CRT Pacing
All-Cause Mortality (participants affected / at risk) | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 0/12

LIMITATIONS AND CAVEATS:
Planned interim evaluation of sample size calculation assumptions showed variability higher than assumed and planned sample size underpowered for assumed difference. Objectives were not analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In most cases, contracts allow investigators to publish study results per the protocol and publication plan following Medtronic's review to determine whether confidential information (CI) is disclosed. Any such CI is deleted prior to publication/presentation. Medtronic may not censor/interfere with the publication except as described. Investigators may not publish any single-site publications until the main multi-site study publication has occurred.